CLINICAL TRIAL: NCT07249398
Title: Examining Influence of Social Media Ads on Black and White Adolescents' Food Choices: Master ClinicalTrials.Gov Protocol for Aim 1 (NCT05380505), Aim 2 (NCT06969638) and Aim 3 (NCT06969651).
Brief Title: Influence of Social Media Ads on Food Choice - Master Protocol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH); New York University (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 20-01796; R01CA248441 (NIH)
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Food Selection; Food Choices; Calorie Consumption
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- (Aim 1) Condition 1: Race Congruent Ads (Experimental): Participants will complete a 15-minute survey in which they will be randomized to view and rate Facebook food ads associated with their condition. Then they will complete a food purchasing task in which they will shop in an online store that will display six food items and six beverages. Finally, they will answer demographic questions (e.g., self-reported height and weight) and view a debriefing summary that describes the full purpose of the study.
  Interventions: Behavioral: Racially Congruent Ads
- (Aim 1) Condition 2: Race Incongruent Ads (Experimental): Participants will complete a 15-minute survey in which they will be randomized to view and rate Facebook food ads associated with their condition. Then they will complete a food purchasing task in which they will shop in an online store that will display six food items and six beverages. Finally, they will answer demographic questions (e.g., self-reported height and weight) and view a debriefing summary that describes the full purpose of the study.
  Interventions: Behavioral: Racially Incongruent Ads
- (Aim 2) Black Many Likes (Experimental): Food ads with many "likes" and featuring Black individuals
  Interventions: Behavioral: Black Ads; Behavioral: Many Likes
- (Aim 2) Black Few Likes (Experimental): Food ads with few "likes" and featuring Black individuals
  Interventions: Behavioral: Black Ads; Behavioral: Few Likes
- (Aim 2) White Many Likes (Experimental): Food ads with many "likes" and featuring White individuals
  Interventions: Behavioral: White Ads; Behavioral: Many Likes
- (Aim 2) White Few Likes (Experimental): Food ads with few "likes" and featuring White individuals
  Interventions: Behavioral: White Ads; Behavioral: Few Likes
- (Aim 3) Block 1: Black-Food (Experimental): Exposure to ads with a Black person featuring a food product
  Interventions: Behavioral: Black Ads
- (Aim 3) Block 2: White-Food (Experimental): Exposure to ads with a White person featuring a food product
  Interventions: Behavioral: White Ads
- (Aim 3) Block 3: Black-Non Food (Experimental): Exposure to ads with a Black person featuring a non-food product
  Interventions: Behavioral: Black-Non Food
- (Aim 3) Block 4: White-Non Food (Experimental): Exposure to ads with a White person featuring a non-food product
  Interventions: Behavioral: White-Non Food
- (Aim 3) Block 5: Food-Many Likes (Experimental): Exposure to ads with many "likes" featuring a food product
  Interventions: Behavioral: Many Likes
- (Aim 3) Block 6: Non Food-Many Likes (Experimental): Exposure to ads with many "likes" featuring a non-food product
  Interventions: Behavioral: Non Food-Many Likes
- (Aim 3) Block 7: Food-Few Likes (Experimental): Exposure to ads with few "likes" featuring a food product
  Interventions: Behavioral: Few Likes
- (Aim 3) Block 8: Non Food-Few Likes (Experimental): Exposure to ads with few "likes" featuring a non-food product
  Interventions: Behavioral: Non Food-Few Likes

INTERVENTIONS:
Behavioral: Racially Congruent Ads — (Aim 1) Facebook food ads that are racially congruent.
  Arms: (Aim 1) Condition 1: Race Congruent Ads
Behavioral: Racially Incongruent Ads — (Aim 1) Facebook food ads that are racially incongruent.
  Arms: (Aim 1) Condition 2: Race Incongruent Ads
Behavioral: Black Ads — (Aim 2 and 3) Food ads that feature Black individuals.
  Arms: (Aim 2) Black Few Likes; (Aim 2) Black Many Likes; (Aim 3) Block 1: Black-Food
Behavioral: White Ads — (Aim 2 and 3) Food ads that feature White individuals.
  Arms: (Aim 2) White Few Likes; (Aim 2) White Many Likes; (Aim 3) Block 2: White-Food
Behavioral: Many Likes — (Aim 2 and 3) Food ads that have many "likes"
  Arms: (Aim 2) Black Many Likes; (Aim 2) White Many Likes; (Aim 3) Block 5: Food-Many Likes
Behavioral: Few Likes — (Aim 2 and 3) Food ads that have few "likes"
  Arms: (Aim 2) Black Few Likes; (Aim 2) White Few Likes; (Aim 3) Block 7: Food-Few Likes
Behavioral: Black-Non Food — (Aim 3) Ads featuring a Black person with a non-food product
  Arms: (Aim 3) Block 3: Black-Non Food
Behavioral: White-Non Food — (Aim 3) Ads featuring a White person with a non-food product
  Arms: (Aim 3) Block 4: White-Non Food
Behavioral: Non Food-Many Likes — (Aim 3) Ads with Many "likes" featuring a non-food product
  Arms: (Aim 3) Block 6: Non Food-Many Likes
Behavioral: Non Food-Few Likes — (Aim 3) Ads with Few "likes" featuring a non-food product
  Arms: (Aim 3) Block 8: Non Food-Few Likes

SUMMARY:
This is a Master ClinicalTrials.gov Protocol for study 20-01796:

Aim 1: Examining Influence of Social Media Ads on Black and White Adolescents' Food Choices - Study 1 (NCT05380505)

Aim 2: A Randomized Trial to Examine the Influence of "Likes" in Social Media Food Ads on Black and White Adolescents' Food Purchases - Study 2 (NCT06969638)

Aim 3: Comparing the Effects of Racial Congruence, "Likes," and Food Images in Social Media Ads on Adolescents' Caloric Intake - Study 3 (NCT06969651)

DETAILED DESCRIPTION:
The overall objective is to determine the extent to which racially congruent Facebook food ads influence adolescents' food purchases and actual caloric intake. The investigators are conducting three randomized controlled trials (RCTs). The first two aims involve 15-minute online surveys in which participants (Black and White adolescents) rate ads then complete a "food purchasing" task through a virtual vending machine. The third trial will involve an in-person, hour long lab study where participants will be shown ads while investigators covertly monitor their eye movements.

ELIGIBILITY:
Inclusion Criteria:

1. be 13-17 years of age;
2. identify as only non-Latino White or only Black/African American;
3. report that they log into Facebook at least once daily; and
4. read and speak English.

Exclusion Criteria:

* Any criteria not met as listed above will bar an adolescent from participating in the study.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3650 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of Calories Purchased | Day 0 (approximately 15 minutes )
  Aim 1 Participants only.
Number of Calories Purchased | Day 0 (approximately 5 minutes)
  Aim 2 Participants only.
Caloric Intake | Day 0 (approximately 60 minutes)
  Aim 3 Participants only. Number of calories consumed during the study protocol.
Visual Attention to Ad Features - First Fixation | Day 0 (approximately 60 minutes)
  Aim 3 Participants only. Measured as time to first fixation to the advertisement.
Visual Attention to Ad Features - Gaze Duration | Day 0 (approximately 60 minutes)
  Aim 3 Participants only. Measured as the gaze duration during the advertisement.
Visual Attention to Ad Features - Number of Fixations | Day 0 (approximately 60 minutes)
  Aim 3 Participants only. Measured as the number of fixations on ad features.

SECONDARY OUTCOMES:
Attitude Toward Ad | Day 0 (approximately 15 minutes )
  Aim 1 Participants only. Attitude will be reported on a Likert scale of 1 to 100 (1 = likeable, 100 = unlikeable). The higher the score, the less likeable the ad is to the participant.
Time Spent Viewing Ad | Day 0 (approximately 15 minutes )
  Aim 1 Participants only.
Attitude Toward Ad | Day 0 (approximately 5 minutes)
  Aim 2 Participants only. Attitude will be reported on a Likert scale of 1 to 100 (1 = likeable, 100 = unlikeable). The higher the score, the less likeable the ad is to the participant.
Engagement with Ads | Day 0 (approximately 5 minutes)
  Aim 2 Participants only. Participants indicate in which ways, if any, they would engage with each ad by answering the following question: "How you would respond if you saw this ad on social media"? [Select all that apply: "Like" [heart icon and other emojis], comment, tag a friend, direct message a friend, re-post, none of the above]). The outcome is measured as the number of participants who indicate they would engage with ads.

CONTACTS AND LOCATIONS:
Overall Officials: Marie A. Bragg, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No